CLINICAL TRIAL: NCT03873597
Title: Efficacy of Physical Activity Tele-coaching to Optimise Daily Physical Activity Levels in Lung Transplant Recipients
Brief Title: Physical Activity Tele-coaching in Lung Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 257479
Record Dates: First submitted 2019-03-05; First posted 2019-03-13 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-02

CONDITIONS: Lung Transplant Recipients
Keywords: tele-coaching; physical activity; lung transplant
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Single centre feasibility, parallel, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-coaching + Usual Care (Experimental): This group will undergo a 12 week physical activity tele-coaching intervention consisting of a step-counter and smartphone application, in addition to usual care. Usual care will also include sessions where behavioural strategies will be implemented to promote a physically active lifestyle.
  Interventions: Behavioral: Tele-coaching + Usual Care
- Usual Care (No Intervention): This group will receive sessions where behavioural strategies will be implemented to promote a physically active lifestyle.

INTERVENTIONS:
Behavioral: Tele-coaching + Usual Care — The tele-coaching intervention will be delivered for 3 months following discharge from hospital. This consists of: 1) An interview discussing motivational issues, favourite daily activities and strategies to become more physically active; 2) a step counter 3) a smart phone with tele-coaching application providing activity goals (daily steps), feedback and educational tips on a daily basis. Patients' targets will be automatically revised on a weekly basis, based on performance in the preceding week; (4) a booklet containing home exercises; (5) weekly activity proposals; (6) tele-phone contacts triggered in the case of non-compliance, failure to transmit data or difficulty to progress.
  Arms: Tele-coaching + Usual Care

SUMMARY:
Lung transplantation is an established treatment for patients with end-stage lung disease. Despite the overall success of the treatment to prolong survival and restore lung function, limitations in exercise capacity in the range of 40-60% of predicted normal values are commonly observed, even up to 1 year following the transplant. These persisting limitations are predominantly owed to skeletal muscle abnormalities including muscle atrophy, weakness and increased fatigability, secondary to prolonged deconditioning

Based on objective accelerometry measurements, lung transplant recipients are markedly inactive in daily life compared to their healthy age-matched counterparts. Locomotor muscle weakness following extended hospital and intensive care unit stay, immunosuppressant medications, and the psychological effects of transplantation contribute to persisting physical inactivity and impaired exercise capacity.

Physical activity is a complex health behaviour that is modified by behavioural change interventions. Such interventions may combine the use of wearable monitors (i.e. step counters) with goal setting to increase daily physical activity. In patients with chronic obstructive pulmonary disease (COPD), use of a semi-automated tele-coaching intervention consisting of a step-counter and smartphone application, in combination with behavioural strategies (identification of barriers, goal setting, self-efficacy, motivation, self-monitoring and feedback) increases both daily physical activity levels and quality of life. However, the effectiveness of tele-coaching to induce meaningful improvements in daily steps to transpire into enhanced post-surgery outcomes and improve recovery is yet to be investigated in lung transplant recipients.

Alongside physical activity promotion, incorporation of behavioural strategies are also important in terms of reversing physical inactivity in patients with chronic lung diseases. These strategies address barriers to physical activity including low self-motivation and self-efficacy, and constitute an important component in the management of chronic diseases to improve long term engagement in activities of daily living.

Accordingly, this study will assess the feasibility and clinical efficacy of physical activity tele-coaching to enhance daily physical activity levels within a population at high risk for post-surgical complications. The intervention combines usual care with tele-coaching, which is designed to embed behavioural change and remote coaching to adhere to simple daily physical activity tasks. Behavioural strategies targeted at improving physical activity levels will be applied to all patients prior to hospital discharge, to promote more active lifestyle choices.

DETAILED DESCRIPTION:
Project Plan

This is a single centre, feasibility, parallel two group, randomised controlled trial. We will investigate the effect of adding 3-months of tele-coaching to usual care (UC) versus UC on daily physical activity levels following lung transplantation.

Planned interventions

Following lung transplantation patients will be randomised to: 1) 3 months of tele-coaching in addition to usual care or 2) usual care. Randomisation will be performed independently, with 1:1 allocation and stratified by functional capacity assessed by the 6-min walk distance immediately prior to hospital discharge. Stratification will ensure that patients in the two groups are matched in terms of post-surgery functional capacity. Additionally, whilst in hospital all patients will receive sessions (1-3) where behavioural strategies will be implemented to promote physical activity.

Semi-automated Tele-coaching

The tele-coaching intervention will last for 3 months and will consist of 1) a one-to-one interview exploring motivational factors, potential physical barriers, preferred and non-preferred activities and strategies to become more active. Patients develop a plan to increase physical activity with the interviewer, based on preferred and achievable activities; 2) a step counter providing direct feedback to the patient; 3) smartphone with tele-coaching application providing an activity goal (daily steps) and feedback on a daily basis. Patients' targets are automatically revised every 7 days based on performance in the preceding week; 4) Booklet containing home exercises, which are available in 3 levels of difficulty and consist of general strengthening and stretching exercises; 5) weekly activity proposals; 6) telephone contacts triggered in the case of failure to transmit data or progress. Patients will be asked to wear the step counter during waking hours and interact with the application on a daily basis.

Whilst on the waiting list and during hospital stay post-surgery patients will be familiarised with the operation of the step counter and will be taught how to monitor their daily activity levels (daily/steps), how to transfer data from the step counter to the smart phone and to the platform and how to follow ques to adjust their daily step goals.

Behavioural strategy sessions

Sessions implementing behavioural strategies to promote physical activity will be administered to all patients. Strategies that will be used include; education on the benefits of physical activity, creating a "pros and cons" list, goal setting, self monitoring and rating achievement/pleasure of physical activities.

Assessments

Whilst on the waiting list patients will be screened for any contraindications and will undertake a 6-minute walk test (6MWT) to assess functional capacity and questionnaires to assess anxiety, depression and health related quality of life (HADS and SF-36). Additionally, patients will be given an accelerometer for 7 days to record daily physical activity levels. Prior to hospital discharge or soon afterwards, the following assessment measures will be undertaken; 6MWT, HADS, SF-36 and daily physical activity levels using an accelerometer. All measures will then be repeated after 3, 6 and 12 months. In addition, a record of hospital admissions and emergency department visits will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for single or double lung transplant with a primary diagnosis of Interstitial Lung Disease, Chronic Obstructive Pulmonary Disease, Cystic Fibrosis, Bronchiectasis or Pulmonary Vascular Disease.
2. Males and females aged 18-70 years.
3. Able to provide informed consent
4. Able to speak and read English.

Exclusion Criteria:

1. Severe post-transplant critical illness neuromyopathy
2. Bilateral diaphragmatic weakness
3. Presence of any other significant disease or disorder which, in the opinion of the investigators, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in daily physical activity | Measured for 1 week pre-transplant, measured for 1 week at randomisation (1-2 months post-transplant), 1 week following the 3 month intervention, 1 week at 6 months post randomisation and 1 week at 12 months post-randomisation.
  The daily number of steps will be measured using a triaxial accelerometer.

SECONDARY OUTCOMES:
Change in hospital anxiety and depression score | Measured pre-transplant, at randomisation (1-2 months post-transplant), post intervention, 6 months and 12 months post randomisation.
  Anxiety and depression symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS) questionnaire. Scale measures for Anxiety and Depression are both out of 21. Scoring is grouped as: Normal= 0-7, Borderline abnormal= 8-10, 11-21= Abnormal.
Change in health-related quality of life | Measured pre-transplant, at randomisation (1-2 months post-transplant), post intervention, 6 months and 12 months post randomisation.
  Health-related quality of life will be assessed using The 36-item Short-Form Health Survey (SF-36).
Time to first hospitalisation and emergency department visit | 12 months
  Time to first hospitalisation and emergency department visit following discharge from lung transplantation.
Adherence to tele-coaching intervention | Information gathered after the 3 month intervention
  Adherence of wearing the step counter and performing the tasks of the smartphone interface
Survival | 12 months
  Survival to 12 months post-transplant
Change in functional capacity | Measured pre-transplant and at randomisation (1-2 months post-transplant).
  Functional capacity will be assessed using the 6 minute walk test.
Patient acceptability | Assessed after the 3 month intervention.
  Patient acceptability of the tele-coaching intervention will be assessed using project tailored validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vogiatzis, PhD, Principal Investigator — Northumbria University
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853